CLINICAL TRIAL: NCT01553799
Title: Use of Ultrasound Technology to Check Proper Placement of Tracheal and Endobronchial Tubes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, A.Eldawlatly, professor of anesthesia, King Saud University
Other Study IDs: UST12
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Focus of Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- US check tube
- US check tube, Endobronchial

SUMMARY:
tracheal and endobronchial misplaced will be checked quickly qith US

ELIGIBILITY:
Inclusion Criteria:

* all general anesthesia with trachea and endobronchial intubation

Exclusion Criteria:

* regional anesthesia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all adult of both sexes
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-04